CLINICAL TRIAL: NCT02757989
Title: Allogeneic Hematopoietic Stem Cell Transplantation in Patients With Low or Intermediate-1 Myelodysplastic Syndrome: A Prospective Multicenter Phase II Study Based on Donor Availability on Behalf of the GFM & SFGM-TC
Brief Title: Allogeneic Hematopoietic Stem Cell Transplantation in Patients With Myelodysplastic Syndrome Low Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: Novartis (Industry); Neovii Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDS-ALLO-RISK; 2015-A00292-47 (Other: IDRCB Number)
Record Dates: First submitted 2016-03-31; First posted 2016-05-02 (Estimated); Last update posted 2024-08-02 (Actual); Status verified 2024-02

CONDITIONS: MDS
Keywords: Low risk MDS; Transplantation
MeSH Terms: interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients with donor (Experimental): Patients with a matched donor (8/8 at molecular level unrelated donor or matched sibling)
  Interventions: Other: transplantation
- Patients without donor (No Intervention): Patients without a matched donor

INTERVENTIONS:
Other: transplantation — allogeneic hematopoietic stem cell transplantation in patients with donor
  Arms: Patients with donor

SUMMARY:
Comparison of survival in patients with or without a matched donor at 36 months

DETAILED DESCRIPTION:
Patients with a matched donor (8/8 at molecular level unrelated donor or matched sibling) received an allogeneic hematopoietic stem cell transplantation.

Patients without a matched donor received the best available treatment. All patients will be followed at least 36 months or until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed consent
2. Classical IPSS intermediate 1 or low myelodysplastic syndrome associated with at least one poor prognosis feature:

   1. Intermediate or higher risk revised IPSS
   2. RBC transfusion dependent anemia and failure to 2 or more lines or therapy (including EPO, Lenalidomide or demethylating agent…)
   3. thrombocytopenia < 20 G/L requiring transfusion
   4. neutropenia < 0.5 G/L associated with severe infection (defined as requiring hospitalization)
3. Patient aged ≥ 18 and < 70 years For young patients, 18-45 years, Fanconi disease and dyskeratosis should be ruled out
4. Patient for whom a transplantation from a matched donor, (8/8 (HLA A, B, C, DRB1) identical at molecular level)unrelated donor or matched sibling), is considered irrespective of donor availability
5. Performance status 0-2 on the Eastern Cooperative Oncology Group (ECOG) Scale (At time of screening)
6. Negative pregnancy and adequate contraception (including in male patients wishing to father), if relevant.
7. Wash-out of at least 30 days since a previous treatment with Vidaza, Lenalidomide, EPO or any other treatment inducing cytopenias.

Exclusion Criteria:

1. MDS classified according to classical IPSS as intermediate 2 or High risk
2. Transformation in Acute myeloid Leukemia (AML)
3. Severe active infection or any other uncontrolled severe condition.
4. Organ dysfunctions including the following

   * Hepatic : total bilirubin > 2 times upper limit of normal (ULN) (except moderate unconjugated hyperbilirubinemia due to intra medullary hemolysis or Gilbert syndrome) , alanine transaminase (ALT) and aspartate transaminase (AST) > 3xULN
   * Symptomatic respiratory chronic failure
   * Symptomatic cardiac failure
   * Renal clearance < 60ml/min
5. Prior malignancy (except in situ cervix carcinoma, limited basal cell carcinoma, or other tumors if not active during the last 3 years)
6. MDS with the following causal germline disease : Fanconi anemia, GATA2 related syndromes and telomere disorders

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
overall survival | 36 months
  comparison of overall survival in patients with or without a matched donor (8/8 unrelated donor or matched sibling) at 36 months

SECONDARY OUTCOMES:
quality of life | 12, 24 and 36 months
  comparison of quality of life in patients with or without a matched donor, quality of life assessed by questionnaire (EORTC version 3) at inclusion, 12, 24 and 36 months
number of patients with complete response at 36 month | 36 months
  comparison between patients with or without a donor for cumulative incidence of complete response at 36 month
number of patients with transformation in AML at 36 month | 36 months
  comparison between patients with or without a donor for cumulative incidence of transformation in AML at 36 month
proportion of patients with iron overload | 16 months
  proportion of patients with iron overload (Serum Ferritin (SF)>1000 ng/mL or Red Blood Cells transfusion>20) at time of inclusion and at 16 month after inclusion for non-transplanted patients and 12 months post-transplant for transplanted patients
evolution of innovative iron markers including Non-transferrin binding iron (NTBI), labile plasmatic Iron (LPI) and Hepcidine | 3 and 16 months
  evolution of innovative iron markers including Non-transferrin binding iron (NTBI), labile plasmatic Iron (LPI) and Hepcidine measured at time of inclusion, at 3 month and 16 month post-inclusion for all patients; In transplanted patients these markers will be measured just before conditioning regimen (J-5), Just before the transplantation (J0), at D7, 30, 100 and 12 month after transplant.
efficiency of chelation | 3 and 16 months
  the effect of chelation will be assessed at 3 month after inclusion for all patient and post transplant by measuring Serum ferritin level
number of patients with adverse events grade III and IV as assessed by CTCAE v4.0 | 36 months
  comparison between patients with or without a donor for number of Grade III and IV toxicities (hematological and non-hematological) recorded according to NCI CTCAE criteria versions 4.0 during the 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie Robin, MD, Principal Investigator — Saint-Louis Hospital, Paris, France
Locations (37):
- France (37):
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - Centre hospitalier Victor Dupouy, Argenteuil
  - CHU Jean Minjoz, Besançon
  - Hôpital Avicenne, Bobigny
  - CHU de Haut Lévèque, Bordeaux
  - CHRU Côte de Nacre, Caen
  - CHU Estaing, Clermont-Ferrand
  - CHSF Gilles de Corbeil, Corbeil-Essonnes
  - Hôpital Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - CH Le Mans, Le Mans
  - Hôpital Saint Vincent de Paul, Lille
  - Hôpital Huriez, Lille
  - Hôpital Dupuytren, Limoges
  - Centre hospitalier Lyon Sud, Lyon
  - GHEF, site de Meaux, Meaux
  - CHRU de Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - CHU de Nîmes, Nîmes
  - Hôpital Saint Louis, Paris
  - Hôpital Pitié Salpétrière, Paris
  - Hôpital Cochin, Paris
  - Hôpital Necker, Paris
  - CH Joffre, Perpignan
  - CHU de Poitiers, Poitiers
  - CH René Dubos, Pontoise
  - CHU de Reims, Reims
  - Hôpital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Curie, Saint-Cloud
  - Institut de cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Hôpital civil, Strasbourg
  - IUCT-Oncopole, Toulouse
  - Hôpital Bretonneau, Tours
  - Hôpital de Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Sebert M, Thepot S, Cluzeau T, Duployez N, Lefebvre T, Chaffaut C, Orvain C, Loschi M, Peterlin P, Chevallier P, D'Aveni M, Rubio MT, Rauzy O, Huynh A, Charbonnier A, Sapena R, Chermat F, Ceballos P, Fossard G, Nguyen S, Park S, Ades L, Peffault de Latour R, Preudhomme C, Fenaux P, Chevret S, Robin M. Transplantation in patients with lower-risk MDS: a prospective phase 2 trial based on donor availability. Blood Adv. 2026 Jan 27;10(2):494-504. doi: 10.1182/bloodadvances.2025017035. PMID 41061188
- [Derived] Robin M, Fenaux P. Which lower risk myelodysplastic syndromes should be treated with allogeneic hematopoietic stem cell transplantation? Leukemia. 2020 Oct;34(10):2552-2560. doi: 10.1038/s41375-020-0967-x. Epub 2020 Jul 13. PMID 32661295